CLINICAL TRIAL: NCT05476978
Title: Utilization of Artificial Intelligence for the Development of an EUS-convolution Neural Network Model Trained to Differentiate Pancreatic Cancer From Other Pancreatic Solid Lesions
Brief Title: Artificial Intelligence in EUS for Diagnosing Pancreatic Solid Lesions
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); LanZhou University (Other)
Responsible Party: Principal Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Other Study IDs: EUS-AI 2022
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatitis, Chronic; Pancreatic Neuroendocrine Tumor; Autoimmune Pancreatitis
Keywords: artificial intelligence; endoscopic ultrasound
MeSH Terms: conditions — Pancreatitis, Chronic; Adenoma, Islet Cell; Autoimmune Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreas-EUS: Patients since 2014 with EUS pictures of normal pancreas or pancreatic solid lesions have been included in this cohort.
  Interventions: Diagnostic Test: EUS-AI model

INTERVENTIONS:
Diagnostic Test: EUS-AI model — The test subset (approximately 20% of total patients) is reserved for the final evaluation of the EUS-AI model. Clinical parameters and EUS pictures of each patient in the test subset will be inputed into the trained EUS-AI model, and the most possible diagnosis will be given by the model.

SUMMARY:
We aim to develop an EUS-AI model which can facilitate clinical diagnosis by analyzing EUS pictures and clinical parameters of patients.

DETAILED DESCRIPTION:
EUS is considered to be a more sensitive modality than CT in detecting pancreatic solid lesions due to its high spatial resolution. However, the diagnostic performance is largely dependent on the experience and the technical abilities of the practitioners. Therefore, we aim to develop an objective EUS diagnostic model based on the convolutional neural network, an artificial intelligence technique. In addition, clinical parameters such as risk factors, tumor biomarkers and radiology findings are also added to this artificial intelligence model in order to mimic the actual clinical diagnosis procedures and to increase the performance of this model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent EUS using a curved line array echoendoscope (GF-UCT260; Olympus Medical Systems) since 2014 in our affiliation.
* For each patient, all available native EUS pictures are included.
* Patients' diagnosis are validated by surgical outcomes or fine-needle aspiration (FNA) findings and have a compatible clinical course with a follow-up period of more than 6 months.

Exclusion Criteria:

* The image is of poor quality.
* The images contain unique marks which can potentially bias the model, such as the biopsy needle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from Tongji Hospital, Tongji Medical College, HUST.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
The model's ability to differentiate pancreatic cancer from other pancreatic solid lesion | After the training process of the EUS-AI model is completed
  Receiver operating characteristic (ROC) analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model.

SECONDARY OUTCOMES:
The model's ability to specify the pancreatic solid lesions such as pancreatic cancer, CP, AIP and NET | After the training process of the EUS-AI model is completed
  Receiver operating characteristic (ROC) analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Cui H, Zhao Y, Xiong S, Feng Y, Li P, Lv Y, Chen Q, Wang R, Xie P, Luo Z, Cheng S, Wang W, Li X, Xiong D, Cao X, Bai S, Yang A, Cheng B. Diagnosing Solid Lesions in the Pancreas With Multimodal Artificial Intelligence: A Randomized Crossover Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2422454. doi: 10.1001/jamanetworkopen.2024.22454. PMID 39028670